CLINICAL TRIAL: NCT04348760
Title: Study of Two Inflammatory Cytokines, BAFF and PAF, and Their Clinical Relevance Before and After a Personalized Nutritional Intervention in IBS Subjects
Brief Title: Study of Inflammatory Markers and Symptom Severity in Personalized Nutritional Intervention in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEK Srl (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019_01_IBS
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: IBS - Irritable Bowel Syndrome; Inflammation
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Subjects were then instructed to avoid the foods highlighted in their personal food profile in certain days of the week, and to assume them in 7 of the 21 meals of the week
  Interventions: Behavioral: Rotation Diet

INTERVENTIONS:
Behavioral: Rotation Diet — Based on the food-specific IgG measurement and relative distribution, a personalized food profile was created for each subject identifying 1 to 3 relevant food groups/nutritional clusters. Subjects were then instructed to avoid the foods highlighted in their personal food profile in certain days of the week, and to assume them in 7 of the 21 meals of the week. No calorie restriction was imposed in the diet.

SUMMARY:
Irritable Bowel Syndrome (IBS) is a widespread disease with variable symptoms that have an important impact on the quality of life. Despite the prevalence of IBS, its etiology and pathophysiology are still to be fully understood, but immune response is known to be involved. In this study, the investigators researched the variation of two specific cytokines, B-cell activating factor (BAFF) and platelet-activating factor (PAF), the levels of food-specific IgG and the symptom severity, using Irritable Bowel Syndrome - Symptom Severity Score (IBS-SSS), following a personalized an unrestricted-calorie diet.

DETAILED DESCRIPTION:
The investigators enrolled 30 subjects with diagnosis of IBS, according to Rome-IV criteria, whose inflammatory markers were measured at baseline and after 6 weeks of dietary intervention. The subjects were monitored in a general practice outpatient setting (GP) and nutritional advice was offered remotely via two telephone sessions with a nutritionist. The researchers investigated the variation of two specific cytokines, B-cell activating factor (BAFF) and platelet-activating factor (PAF), the levels of food-specific IgG and the symptom severity, using Irritable Bowel Syndrome - Symptom Severity Score (IBS-SSS).

Data monitoring was ensured by an external monitor (Hippocrates Research, Genova, Italy).

All data entry was in accordance with GCP protocol, and AE were classified using CTCAE 4.0

ELIGIBILITY:
Inclusion Criteria:

* IBS (according to ROME IV criteria)
* blood analysis within 1yr with CBC, TSHr, ESR, CRP, urine, glucose
* attitude to change dietary habits
* willing to follow study protocol

Exclusion Criteria:

* low BMI (<18.5 kg/m2)
* pregnancy
* restrictive dietary habits (e.g. veganism)
* positive FOBT
* faecal calprotectin >200 mcg/g
* known or recurrent bowel infections
* known or recurrent UTI (>3/yr)
* former diverticulitis
* alcohol abuse
* major concurrent disease (e.g. IBD, coeliac disease, eating disorder,...)
* pharmacological treatment with drugs that alter intestinal motility (e.g. PPI, metformin,...)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
BAFF levels | 6 weeks
  reduction of BAFF levels from baseline
PAF levels | 6 weeks
  reduction of PAF levels from baseline

SECONDARY OUTCOMES:
IBS symptom severity | 6 weeks
  IBS symptom severity score reduction from baseline
BMI | 6 weeks
  BMI reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emiliana Tognon, PhD, Principal Investigator — GEK Srl; Mattia Cappelletti, MD, Principal Investigator — SMA srl; Attilio F Speciani, MD, Study Director — GEK Srl
Locations (1):
- GEK srl, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data that underline the results reported in article, after deidentification (text, tables)
Supporting Information: Study Protocol, CSR
Time Frame: immediately following and for 36 months after publication
Access Criteria: Proposals should be directed to the PI/Sponsor. To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Background] Ng QX, Soh AYS, Loke W, Lim DY, Yeo WS. The role of inflammation in irritable bowel syndrome (IBS). J Inflamm Res. 2018 Sep 21;11:345-349. doi: 10.2147/JIR.S174982. eCollection 2018. PMID 30288077
- [Background] Lied GA, Lillestol K, Valeur J, Berstad A. Intestinal B cell-activating factor: an indicator of non-IgE-mediated hypersensitivity reactions to food? Aliment Pharmacol Ther. 2010 Jul;32(1):66-73. doi: 10.1111/j.1365-2036.2010.04314.x. Epub 2010 Mar 26. PMID 20353497
- [Background] Ligaarden SC, Lydersen S, Farup PG. IgG and IgG4 antibodies in subjects with irritable bowel syndrome: a case control study in the general population. BMC Gastroenterol. 2012 Nov 21;12:166. doi: 10.1186/1471-230X-12-166. PMID 23170971
- [Derived] Cappelletti M, Tognon E, Vona L, Basello K, Costanzi A, Speciani MC, Speciani AF. Food-specific serum IgG and symptom reduction with a personalized, unrestricted-calorie diet of six weeks in Irritable Bowel Syndrome (IBS). Nutr Metab (Lond). 2020 Dec 1;17(1):101. doi: 10.1186/s12986-020-00528-x. PMID 33292297